CLINICAL TRIAL: NCT00004647
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Mexiletine for Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Tennessee (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11702; UTENN-4686
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-03

CONDITIONS: Pain; Diabetic Neuropathies; Paresthesia
Keywords: diabetic neuropathy; disease-related problem/condition; neurologic and psychiatric disorders; pain; rare disease
MeSH Terms: conditions — Pain; Diabetic Neuropathies; Paresthesia; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Mexiletine

INTERVENTIONS:
Drug: mexiletine

SUMMARY:
OBJECTIVES:

I. Assess the efficacy and toxicity of mexiletine in the management of paresthesias and pain in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution.

The first group receives oral mexiletine 3 times a day for 6 weeks. The dose is increased after the first week if there are no side effects.

The second group receives a placebo. Patients cross to the alternate treatment after a 1-week washout.

ELIGIBILITY:
Patients with painful diabetic neuropathy

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 1993-03; Study Completion 1999-02

CONTACTS AND LOCATIONS:
Overall Officials: Tulio Bertorini, Study Chair — University of Tennessee

REFERENCES:
- [Background] Bertorini TE, Alzagatiti BI, Horner LH, et al.: Electrophysiological effects of mexiletine in painful neuropathy. Nerve 21(11): 1576, 1998.